CLINICAL TRIAL: NCT04580836
Title: MRI-Guided Stereotactic Body Radiotherapy for the Treatment of Early Stage Kidney Cancer: A Single Arm Phase II Clinical Trial (MRI-MARK)
Brief Title: MRI-Guided Radiation Therapy for the Treatment of Early-Stage Kidney Cancer, the MRI-MARK Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: A study with 0 ACTUAL Enrollment must have Overall Recruitment Status specified as Withdrawn
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0168; NCI-2020-06739 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0168 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-09-21; First posted 2020-10-09 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2021-11

CONDITIONS: Renal Cell Carcinoma; Stage I Renal Cell Cancer AJCC v8; Stage II Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (MRI-guided SBRT) (Experimental): Patients undergo an MRI scan to check the status and location of the disease, including the motion of the tumor during breathing. Two weeks after MRI, patients undergo SBRT over 1-2 hours on 3 non-consecutive weekdays in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase II trial investigates how well MRI-guided stereotactic body radiation therapy works in treating patients with early-stage kidney cancer. Radiation therapy uses high energy radiation to kill tumor cells and shrink tumors. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. This method of radiation delivery is further refined through the incorporation of a MRI into the radiation machine to create a device known as a MRI linear accelerator. During treatment with MRI linear accelerator, continuous MRI images are obtained to allow for real-time treatment monitoring and the ability to adjust treatment plans if minor deviations in anatomy are noted. Giving MRI-guided stereotactic body radiation therapy may help treat patients with early-stage kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate local control following magnetic resonance imaging (MRI)-guided stereotactic body radiation therapy (SBRT) for primary kidney cancer as defined by no growth by imaging at 24 months following SBRT.

SECONDARY OBJECTIVES:

I. To estimate preservation of renal function and to determine frequency of grade 3+ adverse events following SBRT as per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

II. To characterize tumor and treated kidney changes by multiparametric MRI, including utility of diffusion and perfusion changes in renal cell carcinoma (RCC) prior to and after SBRT as biomarkers of treatment response.

III. To estimate the rate of pathologic complete response as determined by tumor biopsy at 24 months following SBRT.

IV. To estimate rate of no progression by Response Evaluation Criteria in Solid Tumors (RECIST) at 24 months (less than 20% growth in largest tumor dimension as measured by imaging).

V. To estimate the rates of overall survival and distant metastasis. VI. To evaluate economic strain following SBRT for primary kidney cancer. VII. Compare planned total doses to true total doses delivered to the target and adjacent normal structures, to correlate true delivered doses to normal structures to grade 3+ toxicity, and to determine the rate of cases in which the prescribed isodose line failed to cover 100% of the internal gross tumor volume (iGTV).

OUTLINE:

Patients undergo an MRI scan to check the status and location of the disease, including the motion of the tumor during breathing. Two weeks after MRI, patients undergo SBRT over 1-2 hours on 3 non-consecutive weekdays in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3, 6, 12, 18, and 24 months, then every 6 months thereafter until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients may enter the study if they are diagnosed with bilateral kidney cancer, multiple lesions in the same kidney, recurrent kidney cancer, or if they have previous or current history of a separate cancer, given all other inclusion criteria met
* Have a pathologically confirmed diagnosis of renal cell carcinoma (RCC) of any histology
* Be a suboptimal surgical or ablation candidate, as determined by patient's primary urologist at MD Anderson Cancer Center and by multi-disciplinary consensus. At or before the time of enrollment, a note documenting multidisciplinary consensus supporting active treatment will be recorded in the patient's chart
* Tumor stage of T1-T2a (i.e. 10cm or less in greatest dimension)
* Be technically and anatomically appropriate for MRI-guided SBRT, as determined by patient's primary radiation oncologist. Factors considered will include distance between tumor and bowel, tumor movement with respiration as assessed by 4-dimensional (4D) computed tomography (CT) scan, and prior radiotherapy
* Multi-disciplinary consensus that active treatment is warranted
* Have Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Have life expectancy of 2 years or more

Exclusion Criteria:

* An MRI contraindication (i.e. pacemaker, severe claustrophobia, or MRI-incompatible device)
* A pre-treatment estimated glomerular filtration rate < 30 cc/min
* Visceral, nodal, or bony metastatic disease
* Is pregnant or expecting to conceive within the projected duration of the trial at the screening visit

  * Female subject of childbearing potential should have a negative urine or serum pregnancy within 6 weeks prior to study registration up to the first fraction of radiation
  * Note: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Has a diagnosis of active scleroderma, lupus, or other rheumatologic disease which in the opinion of the treating radiation oncologist precludes safe radiation therapy
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Estimated)

PRIMARY OUTCOMES:
Time to progression | at 24 months
  Local control will be defined as no growth (stability or regression) in the largest dimension of the treated tumor by comparison of magnetic resonance imaging (MRI) images at baseline and 24 months following completion of stereotactic body radiation therapy (SBRT). The local control rate will be compared to case-matched data from patients undergoing active surveillance at MD Anderson Cancer Center. In terms of the primary efficacy analysis, the local control will be evaluated along with the 95% confidence interval. For patients who progress earlier than 24 months will be considered as local control failure and will be included in the confidence interval calculation. In addition, we will estimate the probabilities of local control utilizing the Kaplan Meier method with corresponding 95% confidence intervals.

SECONDARY OUTCOMES:
Preservation of renal function | Baseline to 24 months
  Patients will undergo split function renal scans to determine glomerular filtration rate (GFR) at baseline, 12 months, and 24 months. Change in GFR will be reported by diving the difference in GFR at baseline and at the respective follow up visit, by baseline GFR. The change of GFR at follow up visits and baseline will be evaluated by paired t-test. Mixed model will be used to explore the change of GFR over time after taking the within-subject correlation.
Treatment related toxicities | Up to 24 months after completion of SBRT
  The frequency of non-laboratory non-fatigue adverse events will be determined, defined as a grade 3+ event following SBRT, attributed to SBRT, and affecting the ipsilateral kidney or an adjacent organ (contralateral kidney, liver, small bowel, large bowel, stomach, spleen, or nerves) as per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Changes in the imaging of primary tumor and treated kidney | Baseline up to 24 months after completion of SBRT
  Patients will undergo MRI of the abdomen at regular intervals (i.e. at 6, 12, 18, and 24 months) permitting analysis of changes in functional imaging biomarkers evaluating tumor and renal perfusion and diffusion, which can be correlated to clinical outcome and toxicities. Mixed model will be used to explore the change of tumor characteristics over time after taking the within-subject correlation. Multi b-value diffusion-weighted imaging (DWI) derived diffusion and perfusion changes will be evaluated over the course of therapy to assess their utility as predictors of renal insufficiency following therapy.
Pathologic response | At 24 months
  All tumors will be biopsied at baseline. When safe and feasible, patients will undergo re-biopsy at 24 months following SBRT. Viability and percent necrosis will be determined by hematoxylin and eosin (H&E) staining. Other stains such as ki67 may be included. Taking pathologic evaluation as gold standard for no viable tumor cells following SBRT, will correlate tumor biopsy results with local control by imaging. McNemar test will also be used to evaluate the agreement between local control (yes versus [vs] no) and pathologic evaluation (responder vs none). Will also calculate sensitivity and specificity of our primary endpoint of local control (no growth by computed tomography [CT] scan at 24 months).
Progression free survival | At 24 months
  Will estimate no progression Response Evaluation Criteria in Solid Tumors (RECIST) at 24 months (less than 20% growth in largest tumor dimension) along with the 95% confidence interval (CI).
Distant metastasis-free survival | Up to 24 months
  Will estimate the probabilities of patients remaining free from distant metastases utilizing the Kaplan Meier method with corresponding 95% CIs. The log rank test will be used to compare the survival difference between important subgroups (such as tumor categories, etc.). Cox model will be conducted to examine the clinical factor effect on time-to-event variables.
Overall survival | Up to 24 months
  Will estimate the probabilities of patient survival utilizing the Kaplan Meier method with corresponding 95% CIs. The log rank test will be used to compare the survival difference between important subgroups (such as tumor categories, etc.). Cox model will be conducted to examine the clinical factor effect on time-to-event variables.
Economic strain of MRI-guided SBRT | Baseline to 24 months
  Assessed using the validated ENRICH questionnaire. Questionnaire scores will be calculated based on standardized manual associated with the instrument. Incomplete surveys (in the event that a participant declines to answer one or more questions) will still be considered valid and will be used for study purposes. Descriptive statistics will be used to summarize scores of the questionnaire. The distribution of each continuous variable will be summarized by its mean, standard deviation, median, and range. The distribution of each categorical variable will be summarized in terms of its frequencies and percentages. We will compare results at each time point to estimate financial toxicity of treatment. The association between patient clinical factor (such as T-stage or histology result) and clinical measurement (e.g., local control, pathologic response, tumor characteristics by MRI) will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Planned doses | up to 1 month
  Will compare planned doses to true total doses delivered to the target and adjacent normal structures.
Correlation of normal tissue true delivered doses with grade 3+ toxicity | Up to 24 months after completion of SBRT
  Will generate target structure and normal tissue dose volume histograms (DVHs) based on the simulation imaging as per routine treatment planning. Verification MR images will then be obtained immediately prior to each delivered fraction, which may or may not prompt an adaptive plan change. Will use the verification MR images and the delivered plan to generate additional target structure and normal tissue DVHs that will approximate "true" delivered dose. Will generate a cumulative true DVH based on each individual fraction, and compare this to the original planning DVH. Normal tissue toxicity will be assessed in light of both the planned and the true DVH. To assess the impact of intrafraction target and normal structure movement, MR images may also be obtained at specified time intervals during an individual treatment fraction.
Rate of cases in which the prescribed isodose line failed to cover 100% of the internal gross tumor volume (iGTV) | Up to 24 months after completion of SBRT
  The frequency of non-laboratory non-fatigue adverse events will be determined per CTCAE version 5.0. These events will be correlated to the true delivered dose received by the associated organ(s). The number of cases in which the prescribed isodose line failed to cover the entirety of the iGTV will be determined, and correlated to outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Tang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT04580836/ICF_000.pdf